CLINICAL TRIAL: NCT05080829
Title: ABL Mutation Register in Patients With ITK Relapsed or Refractory Chronic Myeloid Leukemia
Brief Title: Myeloid Mutations Register in R/R CML
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Grupo Cooperativo de Hemopatías Malignas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HAL368
Record Dates: First submitted 2021-09-06; First posted 2021-10-18 (Actual); Last update posted 2021-10-18 (Actual); Status verified 2021-10

CONDITIONS: Chronic Myeloid Leukaemia Recurrent; Chronic Myeloid Leukemia, in Relapse
Keywords: chronic myeloid leukemia
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mutation Register (Experimental): Measure of myeloid mutations after detection of relapse or refractoriness to ITK treatment
  Interventions: Diagnostic Test: Myeloid mutations measurement

INTERVENTIONS:
Diagnostic Test: Myeloid mutations measurement — Measure of myeloid mutations by NGS when detection of refractory or relapsed CML is done

SUMMARY:
The aim of the study is to know the percentage of ABL mutations in patients with chronic myeloid leukemia that relapsed or are refractory to tyrosine-kinase inhibitors measured with a myeloid mutations panel by NGS.

ELIGIBILITY:
Inclusion Criteria:

* CML diagnosis by the WHO 2016 criteria
* Failure to reach cytogenetic response of Ph chromosome of 36 to 95% at 3 months or BCR/ABL <10% at 6 months of treatment with TKI
* Progression or relapse of the disease after previous response to treatment with TKI
* Validation of adherence to treatment
* Inform consent

Exclusion Criteria:

* Lack of information to complete the register
* Failure to response achievement due lack of adherence to treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-03-30 (Estimated)

PRIMARY OUTCOMES:
Presence of myeloid mutations by Next Generation Sequence | 1 year
  Detection of positive myeloid mutations at detection of relapse or refractoriness to ITK treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Grupo Cooperativo de Hemopatías Malignas, Huixquilucan, State of Mexico, Mexico

IPD SHARING:
Plan to Share IPD: No